CLINICAL TRIAL: NCT03877393
Title: A 12-week, Randomized, Double-blind, and Placebo-controlled Study Evaluating the Effect of Probiotic Supplementation on the Mental Status, Inflammation, And Intestinal Barrier in Major Depressive Disorder Patients Using Gluten-free or Gluten-containing Diet
Brief Title: The Effect of Probiotic Supplementation on the Mental Status, Inflammation, and Intestinal Barrier in Major Depressive Disorder Patients Using Gluten-free or Gluten-containing Diet
Acronym: SANGUT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lublin (Other)
Collaborators: Sanprobi Sp. z o.o., Sp. k., Szczecin, Poland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS192/2019
Record Dates: First submitted 2019-03-05; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Depressive Disorder, Major; Depression
Keywords: Probiotics; dietary supplements; Diet, Gluten-Free; Inflammation; Gastrointestinal Microbiome; Intestinal mucosal permeability; Gut-brain axis; Gut permeability; EEG functional connectivity; Cortisol; Hypothalamic-pituitary-adrenal axis; Cognitive function
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Inflammation | interventions — Diet, Gluten-Free

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, and placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PRO-GFD (Experimental): Probiotic supplementation + gluten-free diet
  Interventions: Combination Product: Probiotic supplementation + gluten-free diet
- PLA-GFD (Placebo Comparator): Placebo supplementation + gluten-free diet
  Interventions: Combination Product: Placebo supplementation + gluten-free diet
- PRO-GD (Experimental): Probiotic supplementation + gluten-containing diet
  Interventions: Combination Product: Probiotic supplementation + gluten-containing diet
- PLA-GD (Placebo Comparator): Placebo supplementation + gluten-containing diet
  Interventions: Combination Product: Placebo supplementation + gluten-containing diet

INTERVENTIONS:
Combination Product: Probiotic supplementation + gluten-free diet — The probiotic and gluten-free diet group (PRO-GFD) will receive one capsule containing the probiotic mixture powder (Sanprobi Stress; Sanprobi sp. z o.o., sp.k., Szczecin, Poland) in the amount of 3 × 10^9 colony forming units (CFU) per day divided in two equal doses, comprising two bacteria strains: Lactobacillus helveticusRosell®-52, Bifidobacterium longumRosell®-175, and excipients: potato starch, magnesium stearate, and the capsule shell of hydroxypropyl methylcellulose. The participants will be asked to consume supplements before breakfast. The group will follow the elimination diet containing no gluten.
  Arms: PRO-GFD
Combination Product: Placebo supplementation + gluten-free diet — The placebo and gluten-free diet group (PLA-GFD) will receive one capsule containing only the excipients, i.e. maize starch, maltodextrins, and the capsule shell. The participants will be asked to consume supplements before breakfast. The group will follow the elimination diet containing no gluten.
  Arms: PLA-GFD
Combination Product: Probiotic supplementation + gluten-containing diet — The probiotic and gluten-containing diet group (PRO-GD) will receive one capsule containing the probiotic mixture powder (Sanprobi Stress; Sanprobi sp. z o.o., sp.k., Szczecin, Poland) in the amount of 3 × 10^9 colony forming units (CFU) per day divided in two equal doses comprising two bacteria strains: Lactobacillus helveticusRosell®-52, Bifidobacterium longumRosell®-175 and excipients: potato starch, magnesium stearate, and the capsule shell of hydroxypropyl methylcellulose. The participants will be asked to consume supplements before breakfast. The group will stay with their current diet.
  Arms: PRO-GD
Combination Product: Placebo supplementation + gluten-containing diet — The placebo and gluten-containing diet group (PLA-GD) will receive one capsule containing only the excipients, i.e. maize starch, maltodextrins, and the capsule shell. The participants will be asked to consume supplements before breakfast. The group will stay with their current diet.
  Arms: PLA-GD

SUMMARY:
More and more evidence confirms the relationship between the gut-brain-microbiota axis and the symptoms of mood disorders. A potential pathway connecting the intestines and the brain in depression is inflammation. Interventions for reducing inflammation and restoring the integrity of the intestinal mucosa are promising approaches in patients with major depressive disorder (MDD). Gut dysbiosis and the diet containing gluten are potential factors may be factors that negatively affect the communication between intestinal and brain. Gluten has a high immunogenic potential and affinity for the intestinal mucosa layer. In patients with an abnormal reaction to gluten, the elimination diet led to improved mood symptoms. However, the relationship between gluten and depression is still poorly understood. Intestinal microbiota can affect the digestion of gluten and reduce its immunogenic potential. Studies have shown that probiotic supplementation has an anti-inflammatory effect, can lead to changes in intestinal permeability and alleviate the symptoms of depression. This evidence supports the need for co-therapy, including the elimination of gluten and the restoration of intestinal eubiosis to reduce inflammation and modulate the gut-brain-microbiota axis. The objective of the SANGUT study is to determine the impact of interventions concerning the gut-brain-microbiota axis (probiotic supplementation, gluten-free diet and their combination) on the mental state, markers of inflammation and markers of intestinal permeability in adult patients with MDD. The study will last 12 weeks and consist of four visits (V): V0 - Screening (Day 0), V1 - Baseline (up to 1 week after Screening), V2 (six weeks after Baseline), V3 - End of the study (12 weeks after Baseline). The main hypothesis is that probiotic supplementation and/or a gluten-free diet will reduce the symptoms of depression, lower the level of inflammatory markers and favourably affect the integrity of the intestinal mucosal barrier.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients aged 18-60 years old;
2. Signed written Informed Consent Form;
3. Meet the DSM-5 criteria for MDD;
4. Body mass index (BMI) ≥18.5 kg/m2 and ≤30 kg/m2;
5. MADRS (Montgomery-Asberg Depression Scale) total score at screening (V0) and at baseline (V1) of 20 points or more (moderate or severe depression);
6. A willingness and motivation to follow the study protocol.

Exclusion Criteria:

1. Diagnosis of autoimmune, neurological, immunocompromised, thyroid, inflammatory bowel diseases, diabetes, cancers, and/or IgE-dependent allergy;
2. Psychiatric comorbidities (except specific personality disorder) including mental retardation, organic brain dysfunction, or addiction (except nicotine and caffeine);
3. High risk of suicide in the investigator's opinion;
4. An infection one month before the study baseline visit (V1);
5. The use of antibiotics and/or probiotics three months prior to the study;
6. Glucocorticosteroids and/or metformin treatment;
7. Intake of any other drugs which in the investigator' opinion may affect the results of study;
8. Intake of any dietary supplementation (except for vitamin D according to the "Vitamin D supplementation guidelines, 2018") which in the investigator' opinion may affect the results of the study;
9. Changes in a pharmacotherapy and/or psychotherapy of MDD 2 weeks before the trial entry;
10. Electroconvulsive therapy (ECT) 12 months before the trial entry;
11. No specific diet (e.g., elimination, vegan, reduction) and changes in physical activity 4 weeks before the trial entry;
12. Pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
The changes in Montgomery-Åsberg Depression Rating Scale(MADRS) total score to measure the severity of depression symptoms | from the date of randomization until the end of the study up to 12 weeks
  A 10-item questionnaire to measure the severity of depressive symptoms in individuals with mood disorders. The assessment is performed by an experienced clinical psychiatrist. Each item yields a score of 0 to 6 (overall score ranges from 0 to 60). The higher score indicates a higher severity of the depressive episode.
  MADRS cut-off points include:
  * 0 to 6: symptom absent
  * 7 to 19: mild depression
  * 20 to 34: moderate depression
  * more than 34: severe depression
The changes in Beck Depression Inventory (BDI) total score to measure the severity of depression symptoms | from the date of randomization until the end of the study up to 12 weeks
  A 21-item multiple-choice self-report inventory to measure the severity of depression. Each item yields a score of 0 to 3 (overall score ranges from 0 to 63). The higher score indicates more severe depression symptoms.
  BDI cut-off points include:
  * 0 to 9: no/minimal depression
  * 10 to 18: mild depression
  * 19 to 29: moderate depression
  * 30 to 63: severe depression
The changes in Symptom Checklist-90 (SCL-90) total score to measure the severity of psychopathological impairment | from the date of randomization until the end of the study up to 12 weeks
  A 90-item self-reported inventory to evaluate a broad range of psychological problems and symptoms of psychopathology. The SCL-90 measure symptom intensity on nine different subscales: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism. Each item yields a score of 0 to 4 (overall score ranges from 0 to 364). The higher score indicates more severity of symptoms.
The changes in the 36-Item Short Form Survey (SF-36) total score to measure the quality of life | from the date of randomization until the end of the study up to 12 weeks
  A 36-item self-reported survey to evaluate a health status including vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. Raw scores are transforming to 0-100 scale. The higher score indicates a better health state.
The changes in the Perceived Stress Scale (PSS-10) total score to measure the stress levels | from the date of randomization until the end of the study up to 12 weeks
  A 10-item self-reported questionnaire to measure the perception of stress. Each item yields a score of 0 to 4 (overall score ranges from 0 to 40). The higher score indicates higher perceived stress.

SECONDARY OUTCOMES:
Changes in serum levels of high-specific C-reactive protein (hs-CRP) | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of interleukin 6 (Il-6) | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of interleukin 1beta (Il-1beta) | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of tumor necrosis factor alpha (TNF-alpha) | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of anti-tissue transglutaminase (anti-TG2) IgG antibodies | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of anti-gliadin (anti-AGA) IgG antibodies | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of anti-gliadin (anti-AGA) IgA antibodies | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of intestinal fatty acid-binding protein (I-FABP/FABP-2) | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of lipopolysaccharide biding protein (LBP) | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of total cholesterol | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of low-density lipoprotein (LDL) cholesterol | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of high-density lipoprotein (HDL) cholesterol | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of triglycerides (TG) | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of glucose | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of insulin | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of cortisol | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of alanine aminotransferase (ALT) | from the date of randomization until the end of the study up to 12 weeks
Changes in serum levels of aspartate aminotransferase (AST) | from the date of randomization until the end of the study up to 12 weeks
Changes in diversity in microbial community in a single sample (alpha-diversity) | from the date of randomization until the end of the study up to 12 weeks
Changes in diversity in microbial community between samples (beta-diversity) | from the date of randomization until the end of the study up to 12 weeks
Changes in stool short-chain fatty acids (SCFAs) levels | from the date of randomization until the end of the study up to 12 weeks
Changes in electroencephalography (EEG) analysis to assess the functional connectivity (FC) | from the date of randomization until the end of the study up to 12 weeks
  FC will be assessed, based on resting-state EEG-recordings, with the application of a Phase Lag Index (PLI), measuring connectivity strength between a given pair of cortical areas. The global neural network organization will be analyzed with Minimum Spanning Tree algorithm.
Changes in Gastrointestinal Symptom Rating Scale (GSRS) total score to measure intensity of experienced gastrointestinal symptoms | from the date of randomization until the end of the study up to 12 weeks
  A 15-item self-reported questionnaire to measure gastrointestinal symptoms in five clusters: reflux, abdominal pain, indigestion, diarrhoea and constipation. Each item yields a score of 0 to 3 (overall score ranges from 0 to 45). The higher score indicates a higher intensity of experienced symptoms.
Changes in Trail Making Test (TMT) to measure the cognitive abilities | from the date of randomization until the end of the study up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- 1st Department of Psychiatry, Psychotherapy and Early Intervention, Medical University of Lublin, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng QX, Peters C, Ho CYX, Lim DY, Yeo WS. A meta-analysis of the use of probiotics to alleviate depressive symptoms. J Affect Disord. 2018 Mar 1;228:13-19. doi: 10.1016/j.jad.2017.11.063. Epub 2017 Nov 16. PMID 29197739
- [Background] Huang R, Wang K, Hu J. Effect of Probiotics on Depression: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Nutrients. 2016 Aug 6;8(8):483. doi: 10.3390/nu8080483. PMID 27509521
- [Background] Busby E, Bold J, Fellows L, Rostami K. Mood Disorders and Gluten: It's Not All in Your Mind! A Systematic Review with Meta-Analysis. Nutrients. 2018 Nov 8;10(11):1708. doi: 10.3390/nu10111708. PMID 30413036
- [Background] Dinan TG, Cryan JF. Brain-Gut-Microbiota Axis and Mental Health. Psychosom Med. 2017 Oct;79(8):920-926. doi: 10.1097/PSY.0000000000000519. PMID 28806201
- [Background] Dinan TG, Stanton C, Long-Smith C, Kennedy P, Cryan JF, Cowan CSM, Cenit MC, van der Kamp JW, Sanz Y. Feeding melancholic microbes: MyNewGut recommendations on diet and mood. Clin Nutr. 2019 Oct;38(5):1995-2001. doi: 10.1016/j.clnu.2018.11.010. Epub 2018 Nov 17. PMID 30497694
- [Background] Slyepchenko A, Maes M, Jacka FN, Kohler CA, Barichello T, McIntyre RS, Berk M, Grande I, Foster JA, Vieta E, Carvalho AF. Gut Microbiota, Bacterial Translocation, and Interactions with Diet: Pathophysiological Links between Major Depressive Disorder and Non-Communicable Medical Comorbidities. Psychother Psychosom. 2017;86(1):31-46. doi: 10.1159/000448957. Epub 2016 Nov 25. PMID 27884012
- [Background] Karakula-Juchnowicz H, Galecka M, Rog J, Bartnicka A, Lukaszewicz Z, Krukow P, Morylowska-Topolska J, Skonieczna-Zydecka K, Krajka T, Jonak K, Juchnowicz D. The Food-Specific Serum IgG Reactivity in Major Depressive Disorder Patients, Irritable Bowel Syndrome Patients and Healthy Controls. Nutrients. 2018 Apr 28;10(5):548. doi: 10.3390/nu10050548. PMID 29710769
- [Background] Skonieczna-Zydecka K, Marlicz W, Misera A, Koulaouzidis A, Loniewski I. Microbiome-The Missing Link in the Gut-Brain Axis: Focus on Its Role in Gastrointestinal and Mental Health. J Clin Med. 2018 Dec 7;7(12):521. doi: 10.3390/jcm7120521. PMID 30544486
- [Derived] Karakula-Juchnowicz H, Rog J, Juchnowicz D, Loniewski I, Skonieczna-Zydecka K, Krukow P, Futyma-Jedrzejewska M, Kaczmarczyk M. The study evaluating the effect of probiotic supplementation on the mental status, inflammation, and intestinal barrier in major depressive disorder patients using gluten-free or gluten-containing diet (SANGUT study): a 12-week, randomized, double-blind, and placebo-controlled clinical study protocol. Nutr J. 2019 Aug 31;18(1):50. doi: 10.1186/s12937-019-0475-x. PMID 31472678